CLINICAL TRIAL: NCT00828347
Title: A Study of Maintenance Therapy After Intravenous Maxacalcitol for Secondary Hyperparathyroidism
Brief Title: Maintenance Vitamin D Therapy for Secondary Hyperparathyroidism (2HPT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Masataka Adachi, Nephrology KU, Kumamoto University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KumaNeph2
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Results first posted 2016-01-25 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-12

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — alfacalcidol; Hydroxycholecalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1.0 μg/day Alfacalcidol (Other): Alfacalcidol 1.0 μg capsule by mouth, every day for 6 months
  Interventions: Drug: 1.0 μg/day Alfacalcidol
- 0.25 μg/day Alfacalcidol (Other): Alfacalcidol 0.25 μg capsule by mouth, every day for 6 months
  Interventions: Drug: 0.25 μg/day Alfacalcidol

INTERVENTIONS:
Drug: 1.0 μg/day Alfacalcidol — We compared the efficacy of two protocols for maintenance therapy, which were oral administration of alfacalcidol at a dose of 1.0 μg/day in patients whose iPTH level was controlled to < 150 pg/mL by initial maxacalcitol therapy.
  Other Names: One alpha
  Arms: 1.0 μg/day Alfacalcidol
Drug: 0.25 μg/day Alfacalcidol — We compared the efficacy of two protocols for maintenance therapy, which were oral administration of alfacalcidol at a dose of 0.25 μg/day in patients whose iPTH level was controlled to < 150 pg/mL by initial maxacalcitol therapy.
  Other Names: One alpha
  Arms: 0.25 μg/day Alfacalcidol

SUMMARY:
There are still no established protocols for maintenance therapy with intravenous or oral vitamin D preparations after the iPTH target has been achieved.

Therefore, the present study compared the efficacy of two maintenance therapy protocols, i.e., oral administration of alfacalcidol (an oral vitamin D preparation) at a dose of 1.0 ug/day (higher-dose group) or at a dose of 0.25 ug/day (lower-dose group), in patients with secondary hyperparathyroidism who responded to initial maxacalcitol therapy, resulting in the control of iPTH to < 150 pg/mL.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) causes various bone mineral disorders, which have recently been named CKD mineral and bone disorder (CKD-MBD). CKD-MBD presents a spectrum of skeletal abnormalities ranging from high bone turnover state such as osteitis fibrosa, which is seen with SHPT, to states of low bone turnover, which includes osteomalacia and adynamic bone disease. This disease not only increases the risk of cardiovascular disease and mortality, but also increases the risk of fracture. Therefore, it is important to correct the serum inorganic phosphorus (Pi), calcium (Ca) and parathyroid hormone (PTH) levels in dialysis patients, to achieve both appropriate bone turnover and to improve mortality.

The Kidney Disease Outcomes Quality Initiative (K/DOQI) guidelines recommend that the target range of iPTH level for vitamin D therapy should be set at 150-300 pg/mL. In Japan, the mortality risk was significantly lower in the group of patients with iPTH levels < 120 pg/mL than in the standard group set at 180 pg/mL < iPTH < 360 pg/mL, and lowest in the group of patients with 60 pg/mL < iPTH < 120 pg/mL . Based on these findings, Japanese guideline recommend that the target range of iPTH should be set at 60-180 pg/mL .

The efficacies of various oral and intravenous vitamin D preparations for treating SHPT in hemodialysis patients have been reported. and oral or intravenous vitamin D pulse therapy has been clinically applied, especially for patients with severe SHPT.

Up to now, the effectiveness of an oral daily alfacalcidol on SHPT has been confirmed at the dose of 0.25-0.5 μg /day (average 0.364μg /day), 0.5 μg /day, and 1.0 μg /day. The effective dose of OCT has also been verified, and furthermore, it has also been reported that intravenous vitamin D was more effective than oral vitamin D for suppressing PTH secretion. Accordingly, at present intravenous vitamin D therapy is the standard treatment for SHPT, and there are established protocols with regard to dosage and administration. However, no protocols have been established for maintenance therapy using intravenous or oral vitamin D preparations after the control of iPTH target range has been achieved.

Therefore, the present study compared the efficacy of two maintenance therapy protocols for patients with SHPT who responded to initial OCT therapy, resulting in the control of iPTH to <150pg/mL. One was oral administration of alfacalcidol (an oral vitamin D preparation) at a dose of 1.0 μg/day (higher-dose group) and the other was at a dose of 0.25 μg/day (lower-dose group), both of which are clinically effective doses for HD patients with SHPT.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of secondary hyperparathyroidism (iPTH >200 pg/mL to <500 pg/mL)
* Serum Ca < 11.0 mg/dL, and serum P < 7.0 mg/dL.
* At least one year of regular hemodialysis therapy

Exclusion Criteria:

* Patients with a history of hypersensitivity to any ingredient of maxacalcitol
* Patients who had received parathyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Adachi, M.D., Ph.D., Principal Investigator — Department nephrology Kumamoto University
Locations (1):
- Kumamoto University Hospital, Kumamoto, Kumamoto, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Alfacalcidol: oral administration of alfacalcidol at a dose of 1.0 ug/day in patients whose iPTH level was controlled to < 150 pg/mL by initial maxacalcitol therapy.
- Low Dose Alfacalcidol: oral administration of alfacalcidol at a dose of 0.25 ug/day in patients whose iPTH level was controlled to < 150 pg/mL by initial maxacalcitol therapy.
Period: Overall Study
Arm/Group | High Dose Alfacalcidol | Low Dose Alfacalcidol
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Alfacalcidol | Low Dose Alfacalcidol | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.9) | 69.0 (13.7) | 67.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 9 | 5 | 14
Region of Enrollment [Number; unit: participants]
  Japan | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With iPTH Levels Maintained at the Target Levels of 60-180 pg/mL iPTH Level
Time Frame: Participants were followed for 24 weeks
Measure: Number; unit: participants
Arm/Group | High Dose Alfacalcidol | Low Dose Alfacalcidol
Number analyzed (Participants) | 12 | 11
participants
  Controlled cases | 10 | 4
  Uncontrolled cases | 2 | 7
Statistical Analysis 1: Comparison: High Dose Alfacalcidol vs Low Dose Alfacalcidol; Test type: Superiority or Other; p = 0.036, Fisher Exact

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | High Dose Alfacalcidol | Low Dose Alfacalcidol
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
Sample size was small, so it will be necessary to conduct further studies in a larger number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes